CLINICAL TRIAL: NCT02192177
Title: Apoptosis May Have a Role in Etiopathogenesis of Obstetric Cholestasis.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Ali Ozgur Ersoy, Medical Doctor, Zekai Tahir Burak Women's Health Research and Education Hospital
Other Study IDs: M30 Intrahepatic cholestasis
Record Dates: First submitted 2014-07-12; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Pregnancy
Keywords: Apoptosis; intrahepatic cholestasis; obstetric outcomes
MeSH Terms: conditions — Cholestasis, Intrahepatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Maternal venous and umbilical cord blood.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: Pregnant subjects diagnosed with obstetric cholestasis who didn't have any foreknown systemic disease.
- Group 2: entirely healthy pregnant subjects, the control group.

SUMMARY:
Intrahepatic cholestasis of pregnancy is a disease specific to pregnancy period; especially late second and third trimester. We aimed to investigate the role of apoptosis in etiopathogenesis of obstetric cholestasis.

DETAILED DESCRIPTION:
M30 (caspases cleaved Cytokeratin-18 (CK-18) fragment) is a specific apoptosis marker. We aimed to use it to evaluate the apoptotic process.

ELIGIBILITY:
Inclusion Criteria:

* Late second or third trimester of pregnancy.

Exclusion Criteria:

* Foreknown systemic diseases, multiple pregnancy, smoking cigarettes.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who admitted our clinic without foreknown systemic diseases or multiple pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
M30 value as Unit per Liter. | Four months.

SECONDARY OUTCOMES:
Percentage of delivery with cesarean section. | Four months.

CONTACTS AND LOCATIONS:
Overall Officials: Ali O Ersoy, Principal Investigator — Medical doctor
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Ankara, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Del Ben M, Polimeni L, Baratta F, Bartimoccia S, Carnevale R, Loffredo L, Pignatelli P, Violi F, Angelico F. Serum Cytokeratin-18 Is Associated with NOX2-Generated Oxidative Stress in Patients with Nonalcoholic Fatty Liver. Int J Hepatol. 2014;2014:784985. doi: 10.1155/2014/784985. Epub 2014 Jan 29. PMID 24678423
- [Background] Du Q, Zhang Y, Pan Y, Duan T. Lithocholic acid-induced placental tumor necrosis factor-alpha upregulation and syncytiotrophoblast cell apoptosis in intrahepatic cholestasis of pregnancy. Hepatol Res. 2014 May;44(5):532-41. doi: 10.1111/hepr.12150. Epub 2013 May 31. PMID 23627780